CLINICAL TRIAL: NCT07308509
Title: Biomechanical and Developmental Perspectives on Upper Body Postural Adaptations Among School-Aged Children: A Comprehensive Narrative Review
Brief Title: Upper Body Posture Ada[Taion in Children
Status: Completed | Type: Observational
Sponsor: Lincoln University College (Other)
Responsible Party: Principal Investigator, ALZAIDANI ABDULAZIZ ATIAH A, doctor, Lincoln University College
Other Study IDs: LUCMalaysia
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Forward Head Posture; Thoracic Hyperkyphosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: postural instruction — chin in exercise and shoulder retraction

SUMMARY:
Age, body mass index, and modern technological influences predisposed to high prevalence of postural deviations such as forward head posture and thoracic hyperkyphosis, and rounded shoulders among school-aged children. The comprehensive integration of developmental and biomechanical perspectives on these adaptations is limited Upper-body postural adaptations reflect a complex interplay between developmental growth and biomechanical loading. Regular posture assessment in schools and clinical settings is crucial for early detection and culturally tailored prevention. Future longitudinal and cross-cultural studies are essential to establish normative postural values and clarify causal pathways across populations

DETAILED DESCRIPTION:
This review aims to synthesize existing literature addressing age- and BMI-related upper-body postural adaptations and biomechanical loading interact to impact spinal and shoulder alignment, muscular strength, and postural control efficiency in school-aged children.

Methods: A structured narrative synthesis was conducted utilizing literature from PubMed, Scopus, and Google Scholar databases. Inclusion criteria focused on studies involving school-aged children (6-18 years) that investigated head, thoracic, and shoulder posture, as well as muscle strength in relation to age, BMI, and lifestyle factors.

Age-related maturation influences spinal curvature, cervical alignment, and scapular positioning through evolving neuromuscular control. Elevated BMI alters load mechanics and mass distribution, increasing thoracic kyphosis, forward head posture, and shoulder protraction while reducing relative neck and shoulder strength. Obesity-related intramuscular fat infiltration and sedentary life style further impair postural stability and muscle performance

ELIGIBILITY:
Inclusion Criteria:

* school-aged children (6-18 years) has forward head posture, kyphosis and rounded shoulder

Exclusion Criteria:

* systemic disese scoliosis

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: School-aged children (6-18 years) has forward head posture, kyphosis and rounded shoulder
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
forward head posture | one month

CONTACTS AND LOCATIONS:
Locations (1):
- King Faisal Medical Complex, El Taif, El Taif, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided